CLINICAL TRIAL: NCT03778866
Title: Whether the Use of HEPES-buffered Medium Would Affect Live Birth Rate After ICSI
Brief Title: Comparing HEPES-buffered With Bicarbonate-buffered as Handling Media During the ICSI Procedure on Live Birth Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Fawzy (Other Government)
Collaborators: Banoon IVF Center (Other); Quena IVF Center (Unknown)
Responsible Party: Sponsor-Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Organization: Ibn Sina Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IbnSina-HEPES
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bicarbonate-buffered Medium (Experimental)
  Interventions: Other: Bicarbonate-buffered handling medium
- HEPES-MOPS-buffered Medium (No Intervention)

INTERVENTIONS:
Other: Bicarbonate-buffered handling medium — The investigators will evaluate whether the usual bicarbonate culture medium can replace the HEPES buffered medium effectively.
  Arms: Bicarbonate-buffered Medium

SUMMARY:
The pH stability during human gamete handling for intracytoplasmic sperm injection (ICSI) is physiologically sound. As the pH change for bicarbonate-buffered medium, scientists assumed whether the use of HEPES or MOPS buffered medium would provide more stable pH, thereby better outcomes. However, the oil use and time frame outside the incubators have not been accounted for. This study is to evaluate the use of HEPES buffered medium compared with the bicarbonate-buffered medium on ICSI outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ICSI indicated cycles

Exclusion Criteria:

* severe medical illness

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1057 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
live birth rate | 40 weeks
  viable neonate after 30 weeks of Gestation

SECONDARY OUTCOMES:
Clinical pregnancy rate | 12 weeks
  a positive heartbeat on ultrasound at ≥ 7 weeks of gestation
biochemical pregnancy rate | two weeks
  positive b-hCG at ≥ 14 days following embryo transfer
embryo developmental rates | 6 days of culture
  fertilized oocyte per injected ones and developed embryos per fertilized oocytes
Ongoing pregnancy rate | 16 weeks
  Continued pregnancy after week 12 of gestation

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qena Fertility Center, Qina, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, Sohag

IPD SHARING:
Plan to Share IPD: No